CLINICAL TRIAL: NCT06941818
Title: Single Arm, Phase I Clinical Study of HS-IT101 Injection in the Treatment of Advanced Melanoma
Brief Title: HS-IT101 Injection in the Treatment of Advanced Melanoma
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Qingdao Sino-Cell Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-IT101ST01-Ⅰ b
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Advanced Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-IT101 monotherapy (Experimental): TIL Injection administered by intravenous infusion over 30-60 minutes.
  Interventions: Drug: HS-IT101 Injection

INTERVENTIONS:
Drug: HS-IT101 Injection — Adoptive transfer of 5x10^9-6x10^10 autologous TIL to patients i.v. in 30-60 minutes.

SUMMARY:
Single-arm, open-label,interventional study evaluating adoptive cell therapy (ACT) with autologous tumor-infiltrating lymphocyte (TIL) infusion (HS-IT101) after lymphodepletion preparative with fludarabine and cyclophosphamide regimen, followed by IL-2, for the treatment of patients with advanced melanoma.

DETAILED DESCRIPTION:
HS-IT101 is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process, for the treatment of patients with advanced melanoma. The cell transfer therapy used in this study involves patients receiving lymphodepletion treatment with fludarabine and cyclophosphamide, followed by infusion of autologous TIL, then finnaly followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years (inclusive).
2. Histologically or cytologically confirmed advanced, recurrent, or metastatic melanoma (excluding uveal melanoma) that has failed at least one prior line of standard systemic therapy. Subjects with BRAF V600 mutations must have failed BRAF-targeted therapy or been intolerant to such therapy due to toxicity. The necessity and appropriateness of targeted therapy shall be determined by the investigator based on the subject's clinical status.
3. At least one tumor lesion (not subjected to radiotherapy or local therapy within 28 days prior to sampling) must be available for autologous tumor-infiltrating lymphocyte (TIL) preparation, with a minimum tissue weight of ≥0.050 g.
4. At least one measurable lesion (per RECIST 1.1 criteria) must remain after sampling. This lesion must not have received prior radiotherapy or local therapy unless performed >28 days before tumor sampling and demonstrating clear progression.
5. ECOG performance status ≤1.
6. Life expectancy ≥3 months.
7. Adequate organ and bone marrow function at screening, defined as:

   Hematology:

   Absolute neutrophil count (ANC) ≥1.5×10⁹/L; Platelet count (PLT) ≥90×10⁹/L; Hemoglobin (HGB) ≥90 g/L (no transfusion or erythropoietin within 14 days).

   Liver function:

   ALT/AST ≤2.5×ULN (≤5×ULN for liver metastases); Total bilirubin (TBil) ≤1.5×ULN (≤3×ULN if Gilbert's syndrome is confirmed).

   Renal function:

   Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Ccr) ≥60 mL/min (Cockcroft-Gault formula).

   Coagulation:

   Activated partial thromboplastin time (APTT) ≤1.5×ULN; International normalized ratio (INR) and prothrombin time (PT) ≤1.5×ULN.
8. Cardiac function criteria:

   Left ventricular ejection fraction (LVEF) ≥50% by echocardiography; No clinically significant arrhythmias requiring treatment; QTcF interval ≤470 ms (calculated using Fridericia's formula: QTcF = QT/(RR⁰.³³), where RR = 60/heart rate. If initial result is abnormal, repeat twice at 5-minute intervals; use mean value for eligibility); Baseline oxygen saturation >91% in room air.
9. Prior treatment-related toxicities resolved to CTCAE v5.0 Grade ≤1 (excluding alopecia or other toxicities deemed non-risk by the investigator) before tumor sampling.
10. Agreement to use effective non-pharmacologic contraception from informed consent signing until 1 year post-TIL infusion.
11. Willing and able to comply with study visits/procedures, with full understanding of the trial and provision of written informed consent.

Exclusion Criteria:

1. History of severe allergic reactions to medications used in the study (including but not limited to cyclophosphamide, fludarabine, IL-2, gentamicin, amphotericin B, or components of TIL infusion).
2. Uncontrolled clinical conditions, including:

   * Poorly controlled hypertension (resting systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg despite medication);
   * Congestive heart failure (NYHA Class III/IV).
3. Within 6 months prior to screening:

   Deep vein thrombosis, pulmonary embolism, myocardial infarction, severe/unstable arrhythmia, angina pectoris, percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass graft, cerebrovascular accident, transient ischemic attack, or cerebral embolism.
4. Active autoimmune diseases requiring systemic therapy during the study period (except: eczema, vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic treatment in the past 2 years; hypothyroidism managed with thyroid hormone replacement; type 1 diabetes managed with insulin; or autoimmune conditions deemed non-recurrent by the investigator).
5. History of organ transplantation or hematopoietic stem cell transplantation.
6. Use of immunosuppressive drugs (e.g., corticosteroids) within 4 weeks prior to tumor sampling, or concurrent conditions requiring immunosuppressive therapy during the study. Exceptions:

   * Physiological-dose glucocorticoids (≤12 mg/m²/day hydrocortisone or equivalent);
   * Topical or intranasal steroids.
7. Systemic anticancer therapy within 4 weeks prior to preconditioning (including investigational drugs; applies to agents with a half-life <4 weeks [whichever is shorter]) or plans to participate in other interventional trials during the study.
8. Acute/chronic infections, including:

   * HIV positivity, syphilis antibody positivity, or active hepatitis B/C (subjects with HBsAg/HBeAg positivity are eligible if HBV DNA is below the lower limit of detection [LLOD]; HCVAb-positive subjects are eligible if HCV RNA is below LLOD);
   * Active infections requiring systemic therapy or active tuberculosis.
9. Major organ surgery, significant trauma within 4 weeks prior to screening, or planned elective surgery during the trial.
10. Surgical complications or delayed wound healing (investigator-assessed to increase risks of preconditioning, TIL therapy, or IL-2 administration).
11. Other primary malignancies diagnosed within 5 years prior to screening (exceptions: radically treated basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ).
12. Severe respiratory diseases (e.g., interstitial lung disease, severe COPD, pulmonary insufficiency, symptomatic bronchospasm).
13. Gastrointestinal bleeding requiring surgery, intestinal ischemia, or perforation.
14. Leptomeningeal metastasis or uncontrolled/untreated CNS metastases (excludes asymptomatic CNS metastases stable for ≥4 weeks post-treatment without corticosteroids/anticonvulsants).
15. Prior treatment with cell therapy products of the same class.
16. Pregnancy, lactation, or refusal to use contraception.
17. Psychiatric disorders, substance abuse, or other investigator-determined contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | 12 months
  To characterize the safety profile of HS-IT101 in patients with advanced solid tumor as assessed by incidence of adverse events
Serious Adverse Events (SAE) | 12 months
  To characterize the safety profile of HS-IT101 in patients with advanced solid tumor as assessed by incidence of serious adverse events
Objective Response Rate (ORR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor, based on the objective response rate (ORR) as assessed by the Independent Review Committee (IRC) per RECIST v1.1
Time-to-response (TTR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor by assessing the time-to-response (TTR) as assessed by the Investigator per RECIST v1.1
Duration of Response (DOR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor by assessing the duration of response (DOR) as assessed by the Investigator per RECIST v1.1
Disease Control Rate (DCR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor, based on the disease control rate (DCR) as assessed by the Independent Review Committee (IRC) per RECIST v1.1
Progression-Free-Survival (PFS) | Up to 36 months
  To evaluate progression-free-survival (PFS) in patients with advanced solid tumor
Overall Survival (OS) | Up to 36 months
  To evaluate overall survival (OS) in patients with advanced solid tumor

SECONDARY OUTCOMES:
Pharmacokinetic (PK) detection parameters for HS-IT101 | Up to 6 months
  Pharmacokinetic (PK) detection parameters for HS-IT101 injection include peripheral blood lymphocyte subsets and T-cell receptor (TCR) clonality.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No